CLINICAL TRIAL: NCT01051193
Title: A Multicentre, Open-label, Extension Study in Children With Inadequately Controlled Partial Onset Seizures to Investigate Long-term Safety and Tolerability of TRI476 (Oxcarbazepine) as Adjunctive Therapy
Brief Title: Long-term Safety and Tolerability of TRI476 (Oxcarbazepine) in Children With Inadequately Controlled Partial Onset Seizures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRI476B1301E1
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Partial Onset Seizures
Keywords: Seizures; oxcarbazepine; child
MeSH Terms: conditions — Seizures | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRI476 (Experimental): TRI476
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
This study is designed to provide long term safety data of TRI476 in children with inadequately-controlled partial seizures. This study is conducted in patients who complete the core study CTRI476B1301. Blinding is maintained during the transition and dose adjustment phase of the extension study. All patients are treated with TRI476 from the dose adjustment phase onwards. The purpose of study is to confirm that TRI476 as adjunctive therapy is safe.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the double-blind treatment phase of the core study (B1301).
* A parent/legal guardian must be present and give written consent for all patients enrolled in this trial. Patients consent must be obtained using assent document according to patients age.
* Females of childbearing potential must have a negative pregnancy test at Week 8 in the core study B1301.

Exclusion Criteria:

* Patients with medical ineligibility to enter the extension, as assessed by the investigator at each site.
* Patients who participated in the core study, but did not complete it (prematurely discontinued)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (adverse events, laboratory tests, vital signs, electrocardiogram (ECG)) | 52 weeks and until approval/launch

SECONDARY OUTCOMES:
Percent change in the partial seizure frequency per 28 days during the double-blind period from the screening period | 52 weeks and until approval/launch
Seizure Frequency of specific duration | 52 weeks and until approval/launch
Responder rate: defined as the proportion of patients with an at least 50% reduction in the partial epileptic seizure frequency | 52 weeks and until approval/launch
Percent changes in the seizure frequency by subtype | 52 weeks and until approval/launch
Clinical Global Impression of Change | 52 weeks and until approval/launch

CONTACTS AND LOCATIONS:
Locations (24):
- Japan (24):
  - NPC Investigative Site, Nagoya, Aichi-ken
  - NPC Investigative Site, Ōbu, Aichi-ken
  - NPC Investigative Site, Matsuyama, Ehime
  - NPC Investigative Site, Fukuoka, Fukuoka
  - NPC Investigative Site, Kameda-gun, Hokkaido
  - NPC Investigative Site, Sapporo, Hokkaido
  - NPC Investigative Site, Himeji, Hyōgo
  - NPC Investigative Site, Kobe, Hyōgo
  - NPC Investigative Site, Yokohama, Kanagawa
  - NPC Investigative Site, Kōshi, Kumamoto
  - NPC Investigative Site, Kashiwazaki, Niigata
  - NPC Investigative Site, Yufu, Oita Prefecture
  - NPC Investigative Site, Kurashiki, Okayama-ken
  - NPC Investigative Site, Okayama, Okayama-ken
  - NPC Investigative Site, Neyagawa, Osaka
  - NPC Investigative Site, Saitama, Saitama
  - NPC Investigative Site, Moriyama-shi, Shiga
  - NPC Investigative Site, Shizuoka, Shizuoka
  - NPC Investigative Site, Shimotsuke, Tochigi
  - NPC Investigative Site, Bunkyo-ku, Tokyo
  - NPC Investigative Site, Gifu
  - NPC Investigative Site, Niigata
  - NPC Investigative Site, Saitama
  - NPC Investigative Site, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided
NPC is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com